CLINICAL TRIAL: NCT00530543
Title: Effects of Gait Training With Assistance of a Robot-Driven Gait Orthosis in Hemiparetic Patients After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007-01-039
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Stroke
Keywords: Robot; Gait; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Robot-assisted gait training

SUMMARY:
The purpose of this study is to investigate the effects of robot-assisted gait training on active walking in the patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1st-ever-stroke
* hemiplegic patient after stroke
* who can stand independently, but cannot walk more than 10 meters independently
* whose muscle powers of hip and knee are more than poor on manual muscle test

Exclusion Criteria:

* previous gait difficulty before stroke onset
* arthralgia on lower extremity
* uncontrolled hypertension or hypotension
* severe medical illness

Ages: 16 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hoon Jeong, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea